CLINICAL TRIAL: NCT03593954
Title: An Open-Label, Fixed-Sequence Study in Healthy Subjects to Assess the Effect of Ritonavir on the Single-Dose Pharmacokinetics of JNJ-61393215
Brief Title: A Study to Assess the Effect of Ritonavir on the Single-Dose Pharmacokinetics of JNJ-61393215 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108479; 61393215EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-61393215 2 mg + Ritonavir 100 mg (Experimental): Participants will receive suspension of JNJ-61393215 2 mg (Day 1 and 5) orally and tablet of Ritonavir 100 mg twice a Day (Day 4-14) orally.
  Interventions: Drug: JNJ-61393215; Drug: Ritonavir

INTERVENTIONS:
Drug: JNJ-61393215 — Participants will receive 2 oral administrations of 2 mg JNJ-61393215 as oral suspension.
Drug: Ritonavir — Participants will receive 100 mg of ritonavir tablet orally.

SUMMARY:
The primary purpose of this study is to assess the effect of ritonavir, on the single-dose pharmacokinetics (PK) of JNJ-61393215 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants or female participants of non-childbearing potential between 18 and 55 years of age, inclusive
* Before enrollment, female participants must be of non-childbearing potential; postmenopausal state is defined as no menses for 12 months without an alternative medical cause, as documented by medical records or physician's notes and Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy
* Participants must have a body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive (BMI = weight/height^2) and body weight not less than 50 kg
* Participant must be healthy based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and admission to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* Participant has any clinically significant abnormal findings in physical examination, vital signs or 12-lead ECG [including QT corrected according to Fridericia's formula (QTcF) greater than (>) 450 milliseconds (msec) and less than or equal to (=<) 470 (milliseconds) msec for females, Left Bundle Branch Block, atrioventricular (AV) Block second degree or higher, permanent pacemaker or implantable cardioverter defibrillator (ICD)] at screening or admission (up to Day 1 predose), which in the opinion of the investigator are not appropriate and reasonable for the population under study
* Participant has a history of or current liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable
* Participant has any liver function test (including alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP) and bilirubin at screening >1.5 * ULN (upper limit of normal)
* Participant has estimated glomerular filtration rate (eGFR) less than (<) 60 milliliter per minute per 1.73 square meter (mL/min/1.73m^2) at screening (provided by the local laboratory)
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  Cmax is the maximum observed plasma concentration.
Last Quantifiable Plasma Concentration (Clast) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  Clast is the last quantifiable Plasma concentration.
Time to Reach Maximum Plasma Concentration (Tmax) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  Tmax is the time to reach maximum plasma concentration.
Time of the Last Quantifiable Plasma Concentration (Tlast) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  Tlast is the time to last observed quantifiable plasma concentration.
Area Under Plasma-Concentration Time Curve from Time 0 to Time of Last Quantifiable Concentration (AUClast) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  AUClast is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under Plasma-Concentration Curve from Time 0 to Infinite Time (AUCinfinity) of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  AUCinfinity is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
First-Order Rate Constant Associated with the Terminal Portion of the Curve [Lambda(z)] of JNJ-61393215 | Predose; Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hour [h]); Day 2 (24h); Day 3 (48 and 60h); Day 4 (71h 55 minutes); Day 5 (predose, 1, 2, 3, 4, 6, 8, and 16h); days 6 to 14 (Predose); Day 15 (24 h)
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Approximately 8 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA International, Salt Lake City, Utah, United States